CLINICAL TRIAL: NCT05705973
Title: A Post-Market Clinical Follow-up Study With Ultimaster Nagomi™ Sirolimus Eluting Coronary Stent System in Complex PCI Subjects
Brief Title: Ultimaster Nagomi™ Sirolimus Eluting Coronary Stent System in Complex PCI Patients
Acronym: NAGOMI COMPLEX
Status: Active, not recruiting | Type: Observational
Sponsor: Terumo Europe N.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: T137E4
Record Dates: First submitted 2022-12-09; First posted 2023-01-31 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Disease; Coronary Artery Occlusion; Ischemic Heart Disease
Keywords: Percutaneous Coronary Intervention; Complex Bifurcation Lesion
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Occlusion; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultimaster Nagomi™ — The Ultimaster NagomiTM Sirolimus eluting coronary stent system with Rapid Exchange Balloon Delivery System consists of a balloon expandable intra-coronary L605 cobalt chromium (CoCr) stent with abluminal drug eluting coating, that consists of a blend of Sirolimus and Poly(D,L-lactide-co-caprolactone), pre-mounted onto a high pressure, semi-compliant balloon delivery catheter

SUMMARY:
The NAGOMI COMPLEX PMCF (Post-Market Clinical Follow-up) study has been designed to expand the knowledge about outcomes with the Ultimaster Nagomi™ sirolimus eluting coronary stent system (Ultimaster Nagomi™) in complex PCI subjects. The features for a complex PCI are based upon subgroup analysis of earlier published studies.

DETAILED DESCRIPTION:
The study is a prospective, multi-center, post-market, non-interventional, observational, single-arm study. Subjects with an indication for a PCI according to current European Society of Cardiology (ESC) or national guidelines will be treated with the Ultimaster Nagomi™ in accordance with the intended use. The PCI procedure will be per hospital routine including the option, as per physician preference, to assess the functional severity of the lesion, perform intra-coronary imaging, use lesion preparation devices or to perform a staged procedure. Also, post-procedural anti-platelet medication will be per ESC or national guidelines.

The primary endpoint is Target Lesion Failure (TLF) defined as Cardiovascular Death (CD), Target-Vessel related Myocardial Infarction (TV-MI) and Clinically Driven Target Lesion Revascularization (CD-TLR) at 1 year. Secondary endpoints are a broad set of clinical endpoints defined by the Academic Research Consortium-II to fully characterize the performance of the Ultimaster Nagomi™ stent. Clinical events will be adjudicated by an independent Clinical Events Committee (CEC) to ensure a consistent assessment versus the event definitions. The Data Monitoring Committee (DMC) will simultaneously conduct regular review for accumulating data to ensure proper safety data monitoring. Core lab analysis of the baseline angiograms of bifurcation lesions by Quantitative Coronary Angiography (QCA) will be included. Procedural resource data will be collected for health-economic analysis. Subject reported outcomes will be documented using the EQ-5D-5L questionnaire and the Seattle Angina Questionnaire (SAQ) for the assessment of the quality of life and angina status, respectively.

The study will enroll 3,000 patients from European sites. Follow-up will be 2 years, except for subjects in whom no Ultimaster Nagomi™ stent was implanted and subjects that do not meet the inclusion criteria for a complex PCI as ascertained after the index procedure. These subjects will be followed until discharge.

ELIGIBILITY:
General Inclusion Criteria:

1. Age ≥ 18 years
2. Patient has been informed of the nature of the study and agrees to its provisions, has provided written informed consent as approved by the Institutional Review Board/Ethics Committee of the respective clinical site
3. Ischemic heart disease with an indication for a PCI with, if available and per hospital guidelines, Heart Team consensus for a PCI procedure
4. Intention to treat all lesions requiring a PCI with the Ultimaster Nagomi stent

Complex Procedure Inclusion Criteria

Subject meets ≥ 1 of the complex procedure criteria:

1. Multivessel PCI defined as ≥ 2 native coronary arteries and/or venous or arterial bypass grafts treated with a stent
2. ≥ 3 stents implanted
3. ≥ 3 lesions treated
4. Complex bifurcation lesion defined as true bifurcation lesion (Medina 1.1.1, 1.0.1 or 0.1.1) with a side branch diameter ≥ 2.5 mm plus one of the following:

i) side branch disease > 10 mm ii) calcified lesion iii) thrombotic lesion

e) Bifurcation lesion implanted with two stents

f) Total stent length implanted > 60 mm

g) Chronic total occlusion defined as a 100% occlusion with antegrade TIMI 0 flow with at least a 3-month duration

h) Left main stenting (main stem and/or bifurcation)

i) In-stent restenosis

j) Severe calcified lesion with use of atherectomy, lithotripsy or cutting balloon

Exclusion Criteria:

1. Any surgery requiring general anaesthesia, comorbidity or indication likely necessitating the discontinuation of dual anti-platelet therapy before the recommended duration of dual anti-platelet therapy per the ESC or national guidelines
2. Hypersensitivity or contraindication to aspirin, heparin, L605 cobalt-chromium alloy, sirolimus or its structurally related compounds, lactide polymers or caprolactone polymers that cannot be pre-medicated
3. Known contrast sensitivity that cannot be premedicated
4. Pregnant and breastfeeding women
5. Life expectancy < 1 year for any cardiac or non-cardiac cause
6. Participation in another clinical study that has not yet completed its primary endpoint
7. Earlier enrolment in the Nagomi Complex study
8. Unlikely to be available for follow-up during the duration of the study (2 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have signed the informed consent are considered enrolled upon insertion of the first Ultimaster NagomiTM stent is successfully implanted and the complex procedure criteria are confirmed. It is expected that study enrolment will take approximately 1.5 years. Enrolment will be competitive, i.e. enrolment will be closed once the total number of subjects has been reached irrespective of the number of subjects per individual site. Individual sites can not enroll more than 300 subjects.
  The enrolled patient population is expected to be representative for complex patients because of the limited exclusion criteria and the participation of multiple sites from across Europe
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2026-04-29 (Estimated); Study Completion 2027-04-29 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | at 1-year post procedure
  Defined as the composite of cardiovascular death, target-vessel related myocardial infarction and clinically driven target lesion revascularization.

SECONDARY OUTCOMES:
Delivery success | Intraoperative
  Delivery success is defined as an achievement of successful delivery of study stent to the target lesion, expansion of the study stent and withdrawal of the delivery catheter.
Lesion success | Intraoperative
  Lesion success is defined as the attainment of < 30% residual stenosis by visual estimate and/or < 50% (by QCA) using any percutaneous method (if QCA was not available, the visual estimate of diameter stenosis is used).
Device success | Intraoperative
  Device Success is defined as delivery success with the achievement of a final residual diameter stenosis of the target lesion of < 30% by visual assessment and/or < 50% by QCA, using the assigned device only.
Procedure success | during hospitalization, approximately 3 days
  Procedure Success is defined as the achievement of < 30% residual stenosis by visual assessment in all target lesions using any percutaneous method without the occurrence of death, Q wave or WHO defined non-Q wave, or repeat revascularization of the target lesion during the hospital stay.
Target lesion failure (TLF) | at index procedure, 30 days, 6 months, 1 year, and 2 years
  The composite of cardiovascular death, MI (not clearly attributable to a nontarget vessel) and clinically driven Target lesion revascularization (TLR).
Patient oriented composite endpoint (POCE) | at index procedure, 30 days, 6 months, 1 year, and 2 years
  Defined as composite of all-cause mortality, any MI and any coronary revascularization.
Death and subclassifications | at index procedure, 30 days, 6 months, 1 year, and 2 years
  Death may be subclassified as: Cardiovascular death, Noncardiovascular death or Undetermined death.
  Cardiovascular death may include death caused by acute MI, death caused by sudden cardiac death, including unwitnessed, death resulting from heart failure, death caused by stroke, death caused by cardiovascular procedures, death resulting from cardiovascular hemorrhage, death resulting from other cardiovascular cause.
  Noncardiovascular death may include death from malignancy, death resulting from pulmonary causes, death caused by infection (including sepsis), death resulting from gastrointestinal causes, death resulting from accident/trauma, death caused by other noncardiovascular organ failure, death resulting from other.
  Undetermined cause of death is defined as a death not attributable to any other category because of the absence of any relevant source documents.
Myocardial infarction and subclassifications | at index procedure, 30 days, 6 months, 1 year, and 2 years
  Myocardial infarction - Absolute rise in cardiac troponin (from baseline) ≥35 times upper reference limit, plus 1 (or more) of the following criteria:
  * New significant* Q waves or equivalent
  * Flow-limiting angiographic complications
  * New "substantial" loss of myocardium on imaging * Q-wave criteria requires the development of new Q waves ≥40 ms in duration and ≥1 mm deep in voltage in ≥2 contiguous leads.
Revascularization and subclassifications | at index procedure, 30 days, 6 months, 1 year, and 2 years
  Successful revascularization of all lesions with angiographically a diameter stenosis ≥ 50%
Stent thrombosis (ST) and subclassifications | at index procedure, 30 days, 6 months, 1 year, and 2 years
  Definite ST
  Presence of a thrombus that originates in the stent/scaffold or in the segment 5mm prox. or dist. to the stent/scaffold or in a side branch originating from the stented/scaffolded segment & at least 1 of the ff:
  Acute onset of ischemic symptoms at rest New ECG changes suggestive of acute ischemia Typical rise and fall in cardiac biomarkers Or Pathological confirmation of thrombosis Evidence of recent thrombus within the stent/scaffold determined at autopsy Examination of tissue retrieved ff. thrombectomy
  Probable ST Any MI that is related to documented acute ischemia in the territory of the implanted stent/scaffold w/out angiographic confirmation of stent/scaffold thrombosis and in the absence of any other obvious cause.
  Occlusive thrombus Thrombolysis in MI grade 0/1 flow w/in or prox. to a stent/scaffold segment. Nonocclusive thrombus Intracoronary thrombus defined as a noncalcified filling defect or lucency surrounded by contrast material seen in mu
Bleeding (Bleeding Academic Research Consortium (BARC) 3-5) | at index procedure, 30 days, 6 months, 1 year, and 2 years
  Type 3:Clinical, lab, and/or imaging evidence of bleeding w/ specific healthcare provider responses, as below:
  Type 3a Any BT with overt bleeding Overt bleeding plus Hgb drop ≥3 to < 5 g/dL
  Type 3b Overt bleeding plus Hgb drop ≥5 g/dL Cardiac tamponade Bleeding requiring surgical intervention for control Bleeding requiring IV vasoactive drugs
  Type 3c Intracranial hemorrhage
  Type 4:CABG-related bleeding Perioperative intracranial bleeding w/in 48 hr Reoperation after closure of sternotomy for bleeding control Transfusion of ≥5 U whole blood or packed RBC w/in a 48-hr period Chest tube output ≥2 L w/in a 24-hr period
  Type 5:Fatal bleeding
  Bleeding that directly causes death with no other explainable cause. Categorized as:
  Type 5a Probable bleeding that is clinically suspicious as the cause of death, but bleeding is not directly observed and no autopsy or confirmatory imaging.
  Type 5b Definite bleeding that is directly observed (clinical specimen or imaging)
Balance between bleeding (BARC 3-5) and thrombotic event (myocardial infarction and/or stent thrombosis) | at index procedure, 30 days, 6 months, 1 year, and 2 years
  The number of patients with a BARC 3-5 bleeding in comparison to the number of patients with a myocardial infarction and/or a stent thrombosis.
Utilization of cardiovascular health care resources | at index procedure, 30 days, 6 months, 1 year, and 2 years
  Number of devices used during the procedure and use of anti-platelet and anti-thrombotic medication during the follow-up period.
Quality of Life assessment | at baseline, 30 days, 6 months, 1 year, and 2 years
  Quality of Life assessed as per EuroQl five-dimensional (EQ-5D) questionnaire:
  The first part of the questionnaire contain descriptive questions on 5 dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression, each with 5 levels of responses.
  The second part of the questionnaire contains a standard vertical 20-cm visual analog scale that is calibrated from 'the worst health you can imagine' (scored 0) at its base to 'the best health you can imagine' (scored 100) at its apex.
Angina status assessment Seattle Angina Questionnaire (SAQ) | at baseline, 30 days, 6 months, 1 year, and 2 years
  Angina status will be assessed through the Seattle Angina Questionnaire (SAQ).
  The SAQ is a validated disease-specific instrument for assessing the health status of patients with coronary artery disease.
  Scoring: Scores range from 1-100 with higher scores indicating better health
QCA of the index procedure angiogram for a subset of patients with a Complex Bifurcation Lesion (CBL) | procedure
  Luminal dimensions of bifurcation lesions will be measured by off-line quantitative coronary angiography by a central core laboratory.
  The objective of the QCA is to quantitate and express the benefit of the Proximal Optimisation Technique (POT). The POT balloon positioning is of importance in this technique as well as the balloon diameter to obtain optimal stent apposition in the main branch.

CONTACTS AND LOCATIONS:
Locations (52):
- Klinikum Klagenfurt am Wörthersee, Klagenfurt, Austria
- Belgium (8):
  - Imelda Hospital, Bonheiden
  - C.H.U. Charleroi, Charleroi
  - Ziekenhuis Oost-Limburg, Genk
  - Hopital de Jolimont, La Louvière
  - UZ Leuven, Leuven
  - CHR Citadelle, Liège
  - Clinique Saint-Luc Bouge, Namur
  - CHU UCL Mont Godinne Namur, Yvoir
- East Tallinn Central Hospital, Tallinn, Estonia
- France (9):
  - CHU Jean Minjoz, Besançon
  - Hôpital Louis Pradel, Bron
  - Clinique Louis Pasteur, Essey-lès-Nancy
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital Privé Jacques Cartier, Massy
  - Centre Hospitalier Universitaire de Nîmes, Nîmes
  - Clinique Saint-Hilaire, Rouen
  - Hôpital Foch, Suresnes
  - Clinique Pasteur, Toulouse
- Ireland (3):
  - Mater Private Network, Cork
  - Mater Private Hospital, Dublin
  - Galway University Hospital, Galway
- Italy (2):
  - Monzino Cardiology Center, Milan
  - IRCCS Istituto Auxologico Italiano, Milan
- Netherlands (6):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Rijnstate Ziekenhuis, Arnhem
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Catharina Hospital Eindhoven, Eindhoven
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Maasstad Ziekenhuis, Rotterdam
- Uniwersytecki Szpital Kliniczny w Poznaniu Oddział Kardiologii, Poznan, Poland
- Serbia (2):
  - Dedinje Cardiovascular Institute, Belgrade
  - University Clinical Center of Serbia, Belgrade
- Spain (6):
  - Bellvitge University Hospital, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Juan Ramón Jiménez, Huelva
  - Hospital Universitario de León, León
  - Salamanca University Hospital, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
- Sweden (2):
  - Gävle Hospital, Gävle
  - Karolinska University Hospital, Huddinge
- Switzerland (3):
  - Universitätsspital Basel, Basel
  - Luzerner Kantonsspital, Lucerne
  - Istituto Cardiocentro Ticino, Lugano
- United Kingdom (8):
  - Royal Sussex County Hospital, Brighton
  - Lincolnshire Heart Centre Lincoln County Hospital, Lincoln
  - London North West University Healthcare NHS Trus, London
  - Altnagelvin Area Hospital, Londonderry
  - University Hospital of North Midlands, Newcastle
  - Newcastle Freeman Hospital, Newcastle upon Tyne
  - University Hospital Plymouth NHS trust, Plymouth
  - Worcestershire Royal Hospital, Worcester